CLINICAL TRIAL: NCT00412997
Title: A Phase I Dose-escalation Study of LBH589 Administered Orally in Adult Patients With Advanced Solid Tumors or Cutaneous T-cell Lymphoma
Brief Title: LBH589 in Adult Patients With Advanced Solid Tumors or Cutaneous T-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B1101
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Tumors; Cutaneous T-Cell Lymphoma
Keywords: advanced solid tumor; Cutaneous T-cell lymphoma; Phase I; HDAC inhibitor; Adult patients
MeSH Terms: conditions — Neoplasms; Lymphoma, T-Cell, Cutaneous | interventions — Panobinostat

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589
  Other Names: panobinostat

SUMMARY:
The phase I study will evaluate the safety, efficacy and pharmacokinetics of LBH589B in adult patients with advanced solid tumors or Cutaneous T-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Patients with either a) histologically-confirmed, advanced solid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists, or b) cytopathologically confirmed cutaneous T-cell lymphoma (CTCL) whose disease has progressed despite standard therapy or for whom no standard therapy exists. Inclusion is irrespective of stage of disease or extent of prior therapy.
* World Health Organization (WHO) Performance Status of ≤ 2
* Patients must have the adequate laboratory values

Exclusion Criteria:

* Patients with a history of primary CNS tumors
* Patients with any history of brain metastases
* Patients with any peripheral neuropathy ≥ CTCAE grade 2
* Patients with unresolved diarrhea ≥ CTCAE grade 2
* Impairment of cardiac function
* Impairment of gastrointestinal (GI) function or GI disease
* Liver or renal disease

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum-tolerated dose of LBH589 | 1st cycle

SECONDARY OUTCOMES:
Safety and tolerability assessed by AEs, SAEs and laboratory values. | Every 2 weeks
To characterize the pharmacokinetic (PK) profile of LBH589 | every 3 cycles
To assess antitumor activity of LBH589 | every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Tokyo, Japan